CLINICAL TRIAL: NCT02948244
Title: Effect of Creatine Monohydrate on Functional Muscle Strength and Muscle Mass in Children With FSHD: a Multi-centre, Randomised, Double-blind Placebo-controlled Crossover Trial
Brief Title: Effect of Creatine Monohydrate on Functional Muscle Strength in Children With FSHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36298
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Facio-Scapulo-Humeral Dystrophy; FSHD2; FSHD1
Keywords: fshd; creatine monohydrate; children; pediatrics; Facio-Scapulo-Humeral Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Active/Placebo (Active Comparator): Participants will receive 3 months of creatine monohydrate followed by a 6 week washout period followed by 3 months of placebo.
  Interventions: Dietary Supplement: Creatine Monohydrate; Dietary Supplement: Placebo
- Group B - Placebo/Active (Active Comparator): Participants will receive 3 months of placebo followed by a 6 week washout period followed by 3 months of creatine monohydrate.
  Interventions: Dietary Supplement: Creatine Monohydrate; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Synthetically produced dietary supplement Creatine Monohydrate will be used in powder form reconstituted to a drink. The dosage will be 100mg/kg/day up to a maximum of 10 grams daily.
Dietary Supplement: Placebo — Placebo

SUMMARY:
This multi-centre, randomised, double-blind, placebo-controlled crossover trial will compare changes in strength-related motor function following treatment with creatine monohydrate to treatment with placebo, as measured by the Motor Function Measure, from baseline to 12 weeks. Eligible subjects will undergo baseline assessments then will be randomised to either creatine monohydrate therapy or placebo for three months, followed by a six week wash-out period, then crossover to a further three months of therapy with either placebo or creatine. Subjects will undergo clinical assessments and study safety assessments at the beginning and end of each treatment period. The study will begin recruitment in early 2017.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 5 and 18 years inclusive at the time of randomisation;
* Has a confirmed genetic diagnosis of Facioscapulohumeral Muscular Dystrophy (FSHD) types 1 or 2;
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Exclusion Criteria:

* Has clinically significant elevation in plasma creatinine level or unexplained hypertension at screening;
* Has a prior diagnosis of chronic renal failure;
* Has a known hypersensitivity to creatine monohydrate of maltodextrin placebo;
* Patients already taking any medications to increase muscle bulk or strength or concomitant use of regular sodium valproate, corticosteroids of alpha agonists such as salbutamol.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Motor Function Measure for Neuromuscular disease | 3 months
  Composite functional outcome measure

SECONDARY OUTCOMES:
Muscle Magnetic Resonance Imaging | 3 months
Muscle Ultrasound Scan | 3 months
Performance of the Upper Limb Measure | 3 months
ACTIVILIM | 3 Months
PedsQL Neuromuscular | 3 months
FSH-COM | 3 months
  FSHD specific composite measure
FSH-Health Index (Pediatric Version) | 3 months
  Patient reported outcome measure specific for patients with FSHD.
Six Minute Walk Test | 3 months
FSHD Severity Score | 3 months
Quantitative muscle strength testing | 3 months
GPX3 Level | 3 months
  Possible biomarker of disease severity in FSHD
Step Counter | 3 months
  Physical activity measure
Laboratory safety monitoring | 3 months
  bloods and urine safety testing (urea and electrolytes, urine plasma creatine:creatinine ratios)

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Woodcock, MBBS, Principal Investigator — Murdoch Children Research Institute/Royal Children Hospital, Melbourne; Monique M Ryan, Principal Investigator — Murdoch Children Research Institute/Royal Children Hospital, Melbourne
Locations (1):
- The Royal Children's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No